CLINICAL TRIAL: NCT05708248
Title: Effect of Pentoxifylline on Anemia in Hemodialysis Patients: Role of Hypoxia Inducible Factor-2 Alpha
Brief Title: Effect of Pentoxifylline on Anemia in Hemodialysis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, hadeer zakaria, PhD student in Clinical Pharmacy and Pharmacy Practice Department, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MDP.22.10.111
Record Dates: First submitted 2022-12-27; First posted 2023-02-01 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Hemodialysis Complication
MeSH Terms: interventions — Pentoxifylline

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental)
  Interventions: Drug: pentoxifylline
- Group II (No Intervention)

INTERVENTIONS:
Drug: pentoxifylline — 400 mg pentoxifylline tablets twice daily with meals for 6 months
  Arms: Group I

SUMMARY:
The primary goal of this clinical trial is to evaluate the promoting effect of pentoxifylline on anemia correction in hemodialysis patients, and involvement of the hypoxia-inducible factor-2 alpha. While, the secondary aim is to evaluate the effect of pentoxifylline on inflammation, hepcidin and other markers of iron homeostasis in these patients. Participants in this trial will be selected to be age and sex ratio matched and will be randomly assigned into two groups. Patients in group I will receive their regular doses of erythropoietin stimulating agents and other routine treatments plus 400 mg pentoxifylline tablets twice daily with meals for 6 months. While, patients in group II will receive their regular doses of erythropoietin stimulating agents and other routine treatments.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes of HD patients
* Age >20 years
* Patients who have adequate hemodialysis for at least 6 months
* Hb level ≤ 10.5 g/dl

Exclusion Criteria:

* Recently dialyzed patients (less than 6 months)
* Patients with known sensitivity to theophylline or other xanthine derivatives
* Severe iron deficiency with serum ferritin < 100 µg/dL and/or TSAT < 20%
* Planning for pregnancy, pregnancy, or lactation
* Patients with severe liver disease or other organ failure
* Previous renal transplantation, noncompliance with medication or HD prescription, or inability to oral drug administration
* Malignancy within last 3 months

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Variation in Hemoglobin (Hb) levels | 6 months
Variation in Hypoxia inducible factor-2 alpha (HIF-2α) levels | 6 months
Variation in Transforming growth factor β1 (TGF-β1) levels | 6 months
Variation in erythropoietin stimulating agents' (ESAs) doses | 6 months
Variation in ESA resistance index (ESA Dose/kg/Week/Hb) | 6 months

SECONDARY OUTCOMES:
Variation in different inflammatory markers levels | 6 months
  Including levels of C-reactive protein (CRP) and Interleukin 6 (IL-6)
Variation in hepcidin hormone levels | 6 months
Variation in different parameters for iron status evaluation | 6 months
  Including serum levels of ferritin, iron and total iron binding capacity (TIBC)

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University Hospital, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zakaria H, Hamdy NA, Sayed-Ahmed NA, El-Mallah A. Pentoxifylline improves anemia through its novel effect on hypoxia-inducible factor-2 alpha in hemodialysis patients: a randomized, double-blind, placebo-controlled clinical trial. Postgrad Med. 2024 Nov;136(8):847-854. doi: 10.1080/00325481.2024.2426448. Epub 2024 Nov 10. PMID 39499142